CLINICAL TRIAL: NCT06576921
Title: Efficacy and Safety of Serplulimab Combined With Nab-paclitaxel and SOX as Neoadjuvant Treatment for Locally Advanced Gastric Cancer or Adenocarcinoma of Esophagogastric Junction: A Multicenter Randomized Controlled Trial
Brief Title: Efficacy and Safety of Serplulimab Combined With Chemotherapy as Neoadjuvant Treatment for Locally Advanced Gastric Cancer or Adenocarcinoma of Esophagogastric Junction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Tang-Du Hospital (Other); Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-AEG/GC-001
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Stomach Neoplasms; Immune Checkpoint Inhibitors
Keywords: Gastric cancer; Adenocarcinoma of Esophagogastric junction cancer; PD-1 antibody
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; S 1 (combination); Oxaliplatin; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This study employed block randomization to allocate subjects in a 1:1 ratio to either the experimental or control group. To ensure balance in sample size between the groups, the randomization sequence was generated using SAS 9.4 software. The randomization list was generated by an independent statistician and securely stored in a password-protected computer system, with corresponding envelopes prepared.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the study, the subjects, the investigator, the sponsor, and the designees are not aware of the randomized allocation, except in the event of emergency unblinding. During the course of treatment with the study drug, if the investigator determines that the study drug is related to a life-threatening situation of the subject, and the investigator considers that knowing the medication of the subject is conducive to the handling of adverse events, an emergency unblinding is allowed. Two sets of sealed blind envelopes were prepared. In the event of an emergency unblinding, the identification number will be used to open the retained envelope to complete the unblinding process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-P-SOX group (Experimental): Neoadjuvant treatment phase: 1.Serplulimab, 4.5 mg intravenously on day 1; 2.Nap-paclitaxel, 260 mg/m2 intravenously on days 1; 3.Oxaliplatin (OXA), 130mg/ /m2, intravenously on days 1; 4.Tigio (S-1), 40-60 mg orally twice daily on days 1 to 14.
  The above treatments will be administered every 3 weeks for three preoperative cycles. Dose adjustment is not allowed and delayed dosing is allowed.
  Surgery phase: Surgery was scheduled 3 to 4 weeks after completion of the last cycle of neoadjuvant treatment. All surgical procedures are performed according to the guidelines of the Japanese Research Society for the Study of Gastric Cancer.
  Adjuvant treatment phase: Adjuvant treatment started 3 to 8 weeks after surgery. Patients will receive three 3-week cycles of adjuvant treatment with S-P-SOX.
  Interventions: Drug: Serplulimab Combined With Chemotherapy
- P-SOX group (Placebo Comparator): Neoadjuvant treatment phase: 1.Nap-paclitaxel, 260 mg/m2 intravenously on days 1; 2.Oxaliplatin (OXA), 130mg/ /m2, intravenously on days 1; 3.Tigio (S-1), 40-60 mg orally twice daily on days 1 to 14.
  The above treatments will be administered every 3 weeks for three preoperative cycles. Dose adjustment is not allowed and delayed dosing is allowed.
  Surgery phase: Surgery was scheduled 3 to 4 weeks after completion of the last cycle of neoadjuvant treatment. All surgical procedures are performed according to the guidelines of the Japanese Research Society for the Study of Gastric Cancer.
  Adjuvant treatment phase: Adjuvant treatment started 3 to 8 weeks after surgery. Patients will receive three 3-week cycles of adjuvant treatment with P-SOX.
  Interventions: Drug: Placebo combined with Chemotherapy

INTERVENTIONS:
Drug: Serplulimab Combined With Chemotherapy — Serplulimab (Dosage form: Lyophilized powder; Unit dose strength: 4.5 mg; Route of administration: IV infusion; Storage requirements: 2-8℃. Protect from light and freezing.) Nap-paclitaxel (Dosage form: Lyophilized powder; Unit dose strength: 100 mg; Route of administration: IV infusion; Storage requirements: <25℃. Protect from light.) S-1 (Dosage form: Capsule; Unit dose strength: 20 mg; Route of administration: Oral; Storage requirements: 20-30℃. Protect from light.) Oxaliplatin (Dosage form: Lyophilized powder; Unit dose strength: 50 mg; Route of administration: IV infusion; Storage requirements: <25℃. Protect from light.) Surgery: All surgical procedures are performed according to the guidelines of the Japanese Research Society for the Study of Gastric Cancer.
  Other Names: Nap-paclitaxel; S-1; Oxaliplatin; surgery
  Arms: S-P-SOX group
Drug: Placebo combined with Chemotherapy — Placebo (Dosage form: Lyophilized powder; Unit dose strength: 4.5 mg; Route of administration: IV infusion; Storage requirements: 2-8℃. Protect from light and freezing.) Nap-paclitaxel (Dosage form: Lyophilized powder; Unit dose strength: 100 mg; Route of administration: IV infusion; Storage requirements: <25℃. Protect from light.) S-1 (Dosage form: Capsule; Unit dose strength: 20 mg; Route of administration: Oral; Storage requirements: 20-30℃. Protect from light.) Oxaliplatin (Dosage form: Lyophilized powder; Unit dose strength: 50 mg; Route of administration: IV infusion; Storage requirements: <25℃. Protect from light.) Surgery: All surgical procedures are performed according to the guidelines of the Japanese Research Society for the Study of Gastric Cancer.
  Other Names: Nap-paclitaxel; S-1; Oxaliplatin; surgery
  Arms: P-SOX group

SUMMARY:
This is a multicenter, double-blind, randomized, phase 2 trial to investigate the efficacy and safety of serlulimab combined with nab-paclitaxel plus SOX versus nab-paclitaxel plus SOX alone as neoadjuvant treatment for locally advanced GC or AEG.

The goal of this clinical trial is to learn if serlulimab combined with nab-paclitaxel plus SOX as neoadjuvant treatment for locally advanced AEG/GC. It will also learn about the safety of serlulimab combined with nab-paclitaxel plus SOX. The main questions it aims to answer are:

Does serlulimab increase the pCR of participants with locally advanced AEG/GC ? What medical problems do participants have when taking serlulimab? Researchers will compare to a placebo (a look-alike substance that contains no drug) to see if serlulimab combined with nab-paclitaxel plus SOX as neoadjuvant treatment for locally advanced AEG/GC.

Participants will:

Eligible patients were randomly assigned to receive serlulimab (4.5 mg intravenously on day 1) combined with chemotherapy (nap-paclitaxel 260 mg/m2 intravenously on days 1, OXA 130mg/ /m2, intravenously on days 1, and S-1 40 to 60 mg orally twice daily depending on BSA on days 1 to 14) or chemotherapy alone every 3 weeks for 3 preoperative cycles followed by 3 postoperative cycles. All patients will be followed for survival.

DETAILED DESCRIPTION:
Gastric Cancer (GC) is the fifth most common malignancy globally and the third leading cause of cancer death. Half of the world's cases occur in eastern Asia [1], which has the highest mortality rate. According to the latest data released by the National Tumor Registration Center, it is estimated that in 2015, there were 679,000 new cases of gastric cancer in China, and 498,000 deaths, ranking second in both incidence and fatality rate among malignant tumors [2]. The overall prognosis is poor, posing a serious threat to human health.

Environmental and genetic factors play an important role in the development of gastric cancer, with common risk factors including age, male gender, smoking, radiation and family history. Specific risk factors for gastric cancer include Helicobacter pylori infection and dietary factors [3]. Helicobacter pylori (H.pylori) infection often leads to chronic gastritis, gastric atrophy, and then intestinal metaplasia, abnormal hyperplasia and gastric cancer [4-6]. Dietary factors include low intake of fruits and vegetables, high salt, and intake of smoked foods.

Radical surgical resection is still the main treatment for non-metastatic gastric cancer, but the postoperative recurrence and metastasis rate is as high as 40-80%, and the 5-year survival rate is 30-60%[7-8]. The treatment mode of neoadjuvant chemotherapy + surgery + adjuvant chemotherapy (perioperative treatment) is an important part of the comprehensive treatment of gastric cancer at present. A number of studies have proved that compared with surgery alone, this treatment mode can reduce the tumor stage, increase the R0 resection rate, and improve the overall survival, without increasing postoperative complications and mortality. The purpose of neoadjuvant chemotherapy is to reduce tumor load and increase the possibility of R0 resection [9], so as to improve the pathological complete response rate. Neoadjuvant chemotherapy can measure a patient's sensitivity to chemotherapy drugs and therefore predict a patient's response to subsequent chemotherapy. At present, it has been confirmed that pathological complete response rate is correlated with overall survival [10]. On September 28, 2019, at the ESMO Conference , Chinese scholars announced the results of the RESOLVE Phase III study on perioperative treatment of locally advanced gastric cancer [11], adding new evidence-based medical evidence for perioperative treatment of such patients. The RESOLVE study is A three-arm, randomized, multicenter, open-label Phase III trial comparing the efficacy and safety of using XELOX (Group A) or SOX (Group B) after radical D2 surgery versus perioperative use of SOX (group C). Finally, 1022 cases of ITT population were included in the analysis. In the perioperative group (group C), the R0 resection rate (92.88%) and the proportion of D2 lymph node dissection (95.59%) showed an increasing trend. The R0 removal rates of group A and group B were 86.47% and 87.83%, respectively. In patients with locally advanced gastric cancer, SOX chemotherapy during perioperative period improved 3-year disease-free survival (62.02% vs 54.78%, P=0.045, HR=0.79, 95%CI 0.62-0.99) compared with XELOX adjuvant. Results of a multicenter Phase III clinical study in France [12] showed that preoperative neoadjuvant chemotherapy with PF regimen significantly increased R0 resection rate compared with surgery alone (84% vs 73%, P=0.04). For initially treated locally advanced gastroesophageal cancer, XELOX regimen has been proven to be as effective as cisplatin combined with fluorouracil regimen [13]. Results of a Chinese study showed that for patients with advanced gastric cancer, the ORR of neoadjuvant chemotherapy with FOLFOX regimen was 70%[14], and the R0 resection rate was significantly improved compared with surgery alone (86% vs 55%, P=0.011). A study from Japan showed [15] that neoadjuvant chemotherapy with SP protocol is safe and effective for stage II and III gastric cancer with lymph node metastasis, with ORR of 75.5% and R0 removal rate of 87.8%. Chinese researchers have found [16] that SOX neoadjuvant application in advanced gastric cancer has an ORR of 68.5%, and the R0 removal rate is also significantly higher than that of operation alone (81.3%vs 73.5%, P=0.040). The results of the recent FLOT4 study [17] showed that the perioperative regimen of 5-fluorouracil + docetaxel + oxaliplatin + calcium folinate (FLOT) was superior to the perioperative regimen of epirubicin + cisplatin + 5-fluorouracil or capecitabine (ECF/ECX) in terms of R0 removal rate (85% vs 78%). P=0.0162).

At present, the recommended preoperative chemotherapy for gastric cancer mainly includes: Epirubicin combined with Cisplatin and fluorouracil (ECF) and its modification, cisplatin combined with fluorouracil (PF), oxaliplatin combined with capecitabine (XELOX), oxaliplatin combined with fluorouracil (FOLFOX), Cisplatin combined with S-1 (SP), oxaliplatin combined with S-1 (SOX), FLOT (5-fluorouracil + docetaxel + oxaliplatin + calcium folinate).

As a highly heterogeneous malignant tumor, gastric cancer is an extremely complex process in which the immune microenvironment plays an important role, and the inhibitory immune microenvironment and immune escape have received more and more attention. programmed death receptor-1 (PD-1) and programmed death ligand-1 (PD-L1) belong to the B7/CD28 superfamily and are very important negative co-stimulatory molecules discovered in recent years. It can negatively regulate the activity of immune cells [18]. PD-1 is the main immunosuppressive molecule on the surface of T cells and B cells. PD-1 has two ligands, PD-L1 and PD-L2. PD-L1 is widely expressed in activated T cells, B cells, macrophages, dendritic cells, and tumor cells. PD-L1 expressed by tumor cells and PD-1 expressed by tumor Infiltrating Lymphocytes (TILs) (mainly CD8+T cells) bind to activate the PD-1/PD-L1 signaling pathway and inhibit the activation of tumor infiltrating lymphocytes. Reduced T cell reactivity leads to T cell incapacitated, induces T cell apoptosis, provides a suitable microenvironment for the development of tumor cells, mediates tumor immune escape, and promotes tumor growth [19]. Blocking the PD-1/PD-L1 signaling pathway can reverse the tumor immune microenvironment and enhance the endogenous anti-tumor immune effect. PD-L1 is highly expressed in various solid malignant tumors [20-21], including non-small cell lung cancer, melanoma, renal cell carcinoma, prostate cancer, breast cancer, stomach cancer, etc., and its expression level varies according to different tumor types. At present, the relationship between PD-L1 expression and prognosis in gastric cancer is still controversial.

In December 2018, the Phase II trial results of the Asian Attract-04 study [22] were published. The study was designed to explore the safety and efficacy of Nivolumab in combination with SOX (Ticeo and oxaliplatin) or XELOX (capecitabine and oxaliplatin) in first-line treatment of advanced, unresectable, or recurrent gastric/gastroesophageal junctional adenocarcinoma. The randomized ratio was 1:1, and the median OS follow-up was not reached in the FAS population (NR (11.9, NR) and NR (11.2, NR), respectively). Median PFS were 9.7 months (5.8-NR) and 10.6 months (5.6-12.5), respectively. The ORR of Nivolumab combined with SOX was 57.1%, and that of Nivolumab combined with XELOX was 76.5%.

In March 2019, the results of KEYNOTE-059 study [23] Cohort 2 and cohort 3 Phase II clinical trials were published. The study cohort 2 and cohort 3 were designed to explore the safety and efficacy of Pembrolizumab± chemotherapy in first-line treatment of advanced gastric or gastroesophageal junction adenocarcinoma. In cohort 2, 25 patients received Pembrolizumab combined with chemotherapy. All patients had an ORR of 60.0%, including 73.3% ORR in the PD-LI positive group and 37.5% ORR in the PD-LI negative group, with a median OS of 13.8 months (8.6-NR). The median PFS was 6.6 months (5.9-10.6). In cohort 3, 31 PD-L1 positive (CPS≥1) patients who received Pembrolizumab monotherapy had an ORR of 25.8%, a median OS of 20.7 months (9.2-20.7), and a median PFS of 3.3 months.

At the American Society of Clinical Oncology Symposium (ASCO) in June 2019, Merck presented the results of the KEYMAT-062 Phase III study [24], which randomized untreated PD-L1-positive advanced gastric or gastroesophageal junction adenocarcinoma into three groups, group 1 being Pembrolizumab monotherapy (Group P). Pembrolizumab combined with chemotherapy in group 2 (P+C) and placebo combined with chemotherapy in group 3 (C) had primary endpoints of PFS in people with PD-L1 CPS≥1 and OS in people with PD-L1 CPS≥1 and CPS≥10. The results suggest that Pembrolizumab combined with chemotherapy is not superior to chemotherapy for OS and PFS in any population. From the perspective of ORR alone, in patients with CPS≥1, the ORR in group P vs group C vs group P+C was 14.8% vs 37.2% vs 48.6%; In patients with CPS≥10, the ORR in group P vs C vs P+C was 25.0% vs 37.8%vs 52.8%. In terms of safety, the P vs C group had better safety, with the incidence of any grade of AE in the P+C vs C group being 94% vs 92%, and the incidence of grade 3-4 TRAE being 71% vs 68%, with no unexpected adverse events.

On November 5, 2022, at the CSCO Annual Meeting, Professor Huang Jing reported on the research related to the treatment of advanced esophageal cancer with Srulizumab - ASTRO-007: In the whole population, the median PFS in the srulizumab and placebo groups was 5.8 months vs5.3 months (HR=0.60, P < 0.0001), and the median OS was 15.3 months vs 11.8 months (HR=0.68, P=0.0020). Among those with PD-L1 CPS≥10, the median PFS for both groups was 7.1 months vs 5.3 months (HR=0.48, P < 0.0001), and the median OS was 18.6 months vs 13.9 months (HR=0.59, P=0.0082). The study also confirmed the significance of srulizumab combined with chemotherapy in the first-line treatment of advanced esophageal cancer, especially in those with CPS > 10.

In other cancers, such as triple negative breast cancer and head and neck squamous cell carcinoma, Pembrolizumab combined with neoadjuvant chemotherapy has shown promising antitumor activity and clinical efficacy. At present, immunotherapy is also being explored in the perioperative period of gastric cancer, such as the phase III clinical study of KEYKEYNOTE 585 perioperative chemotherapy for gastric cancer combined with or without PD-1 inhibitor, and the clinical study of mFOLFOX combined with PD-1 inhibitor for the treatment of gastroesophageal conjoint adenocarcinoma or gastric adenocarcinoma in perioperative period (NCT03488667), etc. In order to provide a new clinical thinking for the treatment of locally advanced gastric cancer.

This is a multicenter, double-blind, randomized, phase 2 trial to investigate the efficacy and safety of serlulimab combined with nab-paclitaxel plus SOX versus nab-paclitaxel plus SOX alone as neoadjuvant treatment for locally advanced GC or AEG. The goal of this clinical trial is to learn if serlulimab combined with nab-paclitaxel plus SOX as neoadjuvant treatment for locally advanced AEG/GC.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 and younger than 75 years
* Primary GC or AEG (Siewert II/III)confirmed pathologically by endoscopic biopsy
* Clinical stage T3/T4N+M0 disease as assessed by CT/MRI, PET-CT, and laparoscopy, if feasible
* At least one measurable lesion according to the RECIST, version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Surgical treatment after neoadjuvant chemotherapy is planned according to clinical staging criteria.
* Life expectancy of at least 3 months
* Acceptable bone marrow, hepatic, and renal function, including: a)Blood routine examination(No blood transfusion within 14 days; No granulocyte colony-stimulating factor (G-CSF) or other hematopoietic stimulating factors were used): white blood cell count ≥3.5 ×109/L, neutrophils ≥1.5 × 109/L, platelet count >100 × 109/L, and hemoglobin ≥90 g/L; b)Hepatic function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST≤2.5×ULN; total bilirubin (TBIL) ≤1.5×ULN (Gilbert syndrome patients, ≤3×ULN); c)Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Ccr) ≥60mL/ min; d)Coagulation function: activated partial thromboplastin time (APTT), international standardized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
* Written informed consent

Exclusion Criteria:

* Squamous cell carcinoma, adenosquamous cell carcinoma, small cell carcinoma, and undifferentiated gastric cancer were confirmed by pathology
* Positive Her-2 detection (IHC3+ or IHC2+ amplified by FISH detection)
* Prior chemotherapy, radiotherapy, hormone therapy, targeted therapy, or immunotherapy
* Contraindications for surgical treatment or chemotherapy
* Presence of distant metastasis
* History of other malignant disease within the past 5 years, except: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that have been treated radically and have shown no signs of disease for at least 5 years
* Any active or history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy
* History of immunodeficiency diseases, including human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or transplantation
* Severe mental disorder
* Presence of digestive tract obstruction, jaundice, acute infectious diseases, inflammatory bowel disease, Crohn's disease, ulcerative colitis, chronic diarrhea, active tuberculosis
* Immunosuppressive drugs are required for 2 weeks or within 2 weeks or during the study period, excluding the following: a) intranasal, inhaled, topical or topical steroid injections (e.g. intra-articular injections); b) Physiological dose of systemic corticosteroids (≤10mg/ day prednisone or equivalent dose); c) Short-term (≤7 days) use of steroids for the prevention or treatment of non-autoimmune allergic diseases;
* Patients who have undergone major surgery or received live virus vaccine within 4 weeks
* Pregnant or breast-feeding women, subjects who are unwilling to receive effective contraception during treatment and within 6 months after the end of treatment (including male subjects who have the ability to impregnate women and female subjects and their male partners)
* Evidence of bleeding tendency or receiving thrombolytics or anticoagulants
* According to the criteria of the term Common Adverse Events (NCI-CTCAE V5.0), the corresponding symptoms have been diagnosed;
* Hepatitis B or hepatitis C virology tests at the time of screening meet any of the following: a) HBsAg positive and HBV-DNA titer ≥104 copy number /mL or ≥2000IU/mL (hepatitis B carriers should ask researchers for appropriate antiviral treatment); b) Active hepatitis C: HCV antibody positive and HCV-RNA higher than the lower detection limit of the assay;
* Allergic to study drugs
* The investigator believes that the subjects have other conditions that may affect their adherence to the protocol and evaluation of the study indicators, and the subjects are not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 3 weeks after completion of the neoadjuvant treatment phase
  postoperative pathological response according to the Mandard tumor regression grading system (TRG), TRG 1 is pCR.

SECONDARY OUTCOMES:
R0 resection rate | 30 days after completion of the surgery phase
  The tumor was completely removed during the operation, and the cutting edge was also negative when viewed under the microscope, that is, the resection effect was perfect and there were no residual components of the tumor
1 year Progression-free survival rate (PFS) | 1 year
  From the beginning of treatment, patients are able to survive for one year with no probability of disease recurrence.
Adverse event (AE) | 90 days after completion of treatment
  Safety of study drugs according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Morbidity | 30 days after completion of the surgery phase
  Discomfort, dysfunction and other problems caused by surgical injury
Mortality | 30 days after completion of the surgery phase
  Proportion of total deaths among all patients undergoing surgery based on observational follow-up (whether cause of death is causally related to surgery or not)
Hospital stay | 90 days after completion of the surgery phase
  From the first day after surgery to the day before discharge
Overall survival | 3 years
  From randomization to the time of death from any cause.
Disease-free survival | 3 years
  The time from the start of randomization until disease recurrences or patients die due to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hong, Ph.D, Principal Investigator — Xijing Hospital of Digestive Diseases, Xijing Hospital, Air force Medical University, Changlexi ST 15, Shaanxi Province, 710032, China
Locations (4):
- China (4):
  - The fourth hospital of Hebei Medical University, Shijiazhuang, Heibei Province
  - Department of Digestive surgery, Xijing Hospital of Digestive Diseases, Air Force Medical University, Xi' an, China, Xi'an, Shaanxi
  - Department of General Surgery, Tangdu Hospital, Air Force Medical University, Xi'an, Shaanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Van Cutsem E, Sagaert X, Topal B, Haustermans K, Prenen H. Gastric cancer. Lancet. 2016 Nov 26;388(10060):2654-2664. doi: 10.1016/S0140-6736(16)30354-3. Epub 2016 May 5. PMID 27156933
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Karimi P, Islami F, Anandasabapathy S, Freedman ND, Kamangar F. Gastric cancer: descriptive epidemiology, risk factors, screening, and prevention. Cancer Epidemiol Biomarkers Prev. 2014 May;23(5):700-13. doi: 10.1158/1055-9965.EPI-13-1057. Epub 2014 Mar 11. PMID 24618998
- [Result] Murakami TT, Scranton RA, Brown HE, Harris RB, Chen Z, Musuku S, Oren E. Management of Helicobacter Pylori in the United States: Results from a national survey of gastroenterology physicians. Prev Med. 2017 Jul;100:216-222. doi: 10.1016/j.ypmed.2017.04.021. Epub 2017 Apr 27. PMID 28457713
- [Result] Uemura N, Okamoto S, Yamamoto S, Matsumura N, Yamaguchi S, Yamakido M, Taniyama K, Sasaki N, Schlemper RJ. Helicobacter pylori infection and the development of gastric cancer. N Engl J Med. 2001 Sep 13;345(11):784-9. doi: 10.1056/NEJMoa001999. PMID 11556297
- [Result] Plummer M, Franceschi S, Vignat J, Forman D, de Martel C. Global burden of gastric cancer attributable to Helicobacter pylori. Int J Cancer. 2015 Jan 15;136(2):487-90. doi: 10.1002/ijc.28999. Epub 2014 Jun 11. PMID 24889903
- [Result] Brar S, Law C, McLeod R, Helyer L, Swallow C, Paszat L, Seevaratnam R, Cardoso R, Dixon M, Mahar A, Lourenco LG, Yohanathan L, Bocicariu A, Bekaii-Saab T, Chau I, Church N, Coit D, Crane CH, Earle C, Mansfield P, Marcon N, Miner T, Noh SH, Porter G, Posner MC, Prachand V, Sano T, van de Velde C, Wong S, Coburn N; International multidisciplinary expert panel. Defining surgical quality in gastric cancer: a RAND/UCLA appropriateness study. J Am Coll Surg. 2013 Aug;217(2):347-57.e1. doi: 10.1016/j.jamcollsurg.2013.01.067. Epub 2013 May 8. No abstract available. PMID 23664139
- [Result] Smyth EC, Nilsson M, Grabsch HI, van Grieken NC, Lordick F. Gastric cancer. Lancet. 2020 Aug 29;396(10251):635-648. doi: 10.1016/S0140-6736(20)31288-5. PMID 32861308
- [Result] Li Z, Shan F, Wang Y, Zhang Y, Zhang L, Li S, Jia Y, Xue K, Miao R, Li Z, Ji J. Correlation of pathological complete response with survival after neoadjuvant chemotherapy in gastric or gastroesophageal junction cancer treated with radical surgery: A meta-analysis. PLoS One. 2018 Jan 25;13(1):e0189294. doi: 10.1371/journal.pone.0189294. eCollection 2018. PMID 29370182
- [Result] Ychou M, Boige V, Pignon JP, Conroy T, Bouche O, Lebreton G, Ducourtieux M, Bedenne L, Fabre JM, Saint-Aubert B, Geneve J, Lasser P, Rougier P. Perioperative chemotherapy compared with surgery alone for resectable gastroesophageal adenocarcinoma: an FNCLCC and FFCD multicenter phase III trial. J Clin Oncol. 2011 May 1;29(13):1715-21. doi: 10.1200/JCO.2010.33.0597. Epub 2011 Mar 28. PMID 21444866
- [Result] Sumpter K, Harper-Wynne C, Cunningham D, Rao S, Tebbutt N, Norman AR, Ward C, Iveson T, Nicolson M, Hickish T, Hill M, Oates J. Report of two protocol planned interim analyses in a randomised multicentre phase III study comparing capecitabine with fluorouracil and oxaliplatin with cisplatin in patients with advanced oesophagogastric cancer receiving ECF. Br J Cancer. 2005 Jun 6;92(11):1976-83. doi: 10.1038/sj.bjc.6602572. PMID 15928658
- [Result] Li ZY, Koh CE, Bu ZD, Wu AW, Zhang LH, Wu XJ, Wu Q, Zong XL, Ren H, Tang L, Zhang XP, Li JY, Hu Y, Shen L, Ji JF. Neoadjuvant chemotherapy with FOLFOX: improved outcomes in Chinese patients with locally advanced gastric cancer. J Surg Oncol. 2012 Jun 15;105(8):793-9. doi: 10.1002/jso.23009. Epub 2011 Dec 20. PMID 22189752
- [Result] Kochi M, Fujii M, Kanamori N, Mihara Y, Funada T, Tamegai H, Watanabe M, Takayama Y, Suda H, Takayama T. Phase II Study of Neoadjuvant Chemotherapy With S-1 and CDDP in Patients With Lymph Node Metastatic Stage II or III Gastric Cancer. Am J Clin Oncol. 2017 Feb;40(1):17-21. doi: 10.1097/COC.0000000000000058. PMID 24662266
- [Result] Li T, Chen L. [Efficacy and safety of SOX regimen as neoadjuvant chemotherapy for advanced gastric cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2011 Feb;14(2):104-6. Chinese. PMID 21365500
- [Result] Dong H, Zhu G, Tamada K, Chen L. B7-H1, a third member of the B7 family, co-stimulates T-cell proliferation and interleukin-10 secretion. Nat Med. 1999 Dec;5(12):1365-9. doi: 10.1038/70932. PMID 10581077
- [Result] Lote H, Cafferkey C, Chau I. PD-1 and PD-L1 blockade in gastrointestinal malignancies. Cancer Treat Rev. 2015 Dec;41(10):893-903. doi: 10.1016/j.ctrv.2015.09.004. Epub 2015 Sep 21. PMID 26412280
- [Result] Sun S, Fei X, Mao Y, Wang X, Garfield DH, Huang O, Wang J, Yuan F, Sun L, Yu Q, Jin X, Wang J, Shen K. PD-1(+) immune cell infiltration inversely correlates with survival of operable breast cancer patients. Cancer Immunol Immunother. 2014 Apr;63(4):395-406. doi: 10.1007/s00262-014-1519-x. Epub 2014 Feb 11. PMID 24514954
- [Result] Hawkes EA, Grigg A, Chong G. Programmed cell death-1 inhibition in lymphoma. Lancet Oncol. 2015 May;16(5):e234-45. doi: 10.1016/S1470-2045(15)70103-8. PMID 25943068
- [Result] Boku N, Ryu MH, Kato K, Chung HC, Minashi K, Lee KW, Cho H, Kang WK, Komatsu Y, Tsuda M, Yamaguchi K, Hara H, Fumita S, Azuma M, Chen LT, Kang YK. Safety and efficacy of nivolumab in combination with S-1/capecitabine plus oxaliplatin in patients with previously untreated, unresectable, advanced, or recurrent gastric/gastroesophageal junction cancer: interim results of a randomized, phase II trial (ATTRACTION-4). Ann Oncol. 2019 Feb 1;30(2):250-258. doi: 10.1093/annonc/mdy540. PMID 30566590
- [Result] Bang YJ, Kang YK, Catenacci DV, Muro K, Fuchs CS, Geva R, Hara H, Golan T, Garrido M, Jalal SI, Borg C, Doi T, Yoon HH, Savage MJ, Wang J, Dalal RP, Shah S, Wainberg ZA, Chung HC. Pembrolizumab alone or in combination with chemotherapy as first-line therapy for patients with advanced gastric or gastroesophageal junction adenocarcinoma: results from the phase II nonrandomized KEYNOTE-059 study. Gastric Cancer. 2019 Jul;22(4):828-837. doi: 10.1007/s10120-018-00909-5. Epub 2019 Mar 25. PMID 30911859
- [Result] Chen DS, Mellman I. Elements of cancer immunity and the cancer-immune set point. Nature. 2017 Jan 18;541(7637):321-330. doi: 10.1038/nature21349. PMID 28102259
- [Result] Zheng C, Zheng L, Yoo JK, Guo H, Zhang Y, Guo X, Kang B, Hu R, Huang JY, Zhang Q, Liu Z, Dong M, Hu X, Ouyang W, Peng J, Zhang Z. Landscape of Infiltrating T Cells in Liver Cancer Revealed by Single-Cell Sequencing. Cell. 2017 Jun 15;169(7):1342-1356.e16. doi: 10.1016/j.cell.2017.05.035. PMID 28622514
- [Result] Azizi E, Carr AJ, Plitas G, Cornish AE, Konopacki C, Prabhakaran S, Nainys J, Wu K, Kiseliovas V, Setty M, Choi K, Fromme RM, Dao P, McKenney PT, Wasti RC, Kadaveru K, Mazutis L, Rudensky AY, Pe'er D. Single-Cell Map of Diverse Immune Phenotypes in the Breast Tumor Microenvironment. Cell. 2018 Aug 23;174(5):1293-1308.e36. doi: 10.1016/j.cell.2018.05.060. Epub 2018 Jun 28. PMID 29961579
- [Result] Zhang L, Yu X, Zheng L, Zhang Y, Li Y, Fang Q, Gao R, Kang B, Zhang Q, Huang JY, Konno H, Guo X, Ye Y, Gao S, Wang S, Hu X, Ren X, Shen Z, Ouyang W, Zhang Z. Lineage tracking reveals dynamic relationships of T cells in colorectal cancer. Nature. 2018 Dec;564(7735):268-272. doi: 10.1038/s41586-018-0694-x. Epub 2018 Oct 29. PMID 30479382

DOCUMENTS (2):
  • Study Protocol (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT06576921/Prot_000.pdf
  • Informed Consent Form (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT06576921/ICF_001.pdf